CLINICAL TRIAL: NCT04564560
Title: Graft Thrombosis After Endovascular Aortic Repair - a Single Center Experience With the Cook Zenith Alpha Spiral-Z®
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 137828
Record Dates: First submitted 2020-09-22; First posted 2020-09-25 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Aorta Aneurysm
Keywords: Stents; Thrombosis
MeSH Terms: conditions — Aortic Aneurysm; Thrombosis | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with Zenith Alpha Spiral-Z®: Patients that from January 2017 until December 2019 received endovascular aortic repair with the Zenith Alpha Spiral-Z® at St. Olavs Hospital
  Interventions: Procedure: Endovascular aortic repair with Zenith Alpha Spiral-Z®

INTERVENTIONS:
Procedure: Endovascular aortic repair with Zenith Alpha Spiral-Z® — The Zenith Alpha Spiral-Z® stent graft may have an increased risk of thrombosis. The intervention in this study is to assess the extent and degree of thrombosis in patients treated with the Zenith Alpha Spiral-Z® during endovascular repair of aortic aneurysm

SUMMARY:
The purpose of this study is to assess the extent of thrombosis in the Zenith Alpha Spiral-Z® stent graft.

DETAILED DESCRIPTION:
Cook Medical has reported thrombus formation with or without occlusion of the Zenith Alpha Spiral-Z®. The purpose of this study is to measure the extent of thrombus formation and occlusion of these stent graft limbs in patients with aortic aneurysms treated at St. Olavs Hospital in 2017, 2018 and 2019. Information is collected from the Norwegian registry for vascular surgery (NORKAR), electronic patient journal and the picture archiving and communication system (PACS). The total number of included patients is estimated to be approximately 100.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have received endovascular treatment with the Zenith Alpha Spiral-Z® for an aortic aneurysm
* The endovascular procedure was performed at St Olavs Hospital from January 2017 until December 2019

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patient treated at St. Olavs Hospital in the period January 2017 until December 2019 with endovascular aortic repair using the Zenith Alpha Spiral-Z® .
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who have got treated post-surgery due to thrombosis or occlusion of stent graft leg | 12-36 months
  Any endovascular or surgical procedure to treat thrombosis or occlusion
Percentage of patients who got an amputation post-surgery due to thrombosis or occlusion of stent graft leg | 12-36 months
  Any amputation in the affected limb / same side as thrombosed stent graft leg
Percentage of patients who died post-surgery | 12-36 months
  Death of any cause during the observation time

CONTACTS AND LOCATIONS:
Overall Officials: Morten Troøyen, md, Study Director — St Olavs Hospital, Dept Radiology and Nuclear Medicine; Birger H Endreseth, md, Study Director — St Olavs Hospital, Dept Surgery
Locations (1):
- St Olavs Hospital, Clinic of Surgery, Clinic of Radiology and Nuclear Medicine, Trondheim, Norway